CLINICAL TRIAL: NCT06295705
Title: Exploring the Effectiveness of Dance as an Intervention to Promote Social-Emotional Health Within the Everyday Lives of Children With ASD
Brief Title: Exploring the Effectiveness of Dance as an Intervention to Promote Social-Emotional Health in Children With Autism Spectrum Disorder (ASD)
Acronym: ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5230588
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hip-Hop Dance (Experimental): The program will be a 7-week occupational therapy led dance program utilizing hip-hop dance as an intervention. Subjects with ASD will dance for 1 time a week for 60 minutes, ending with a dance showcase on the final week.
  Interventions: Behavioral: Hip-Hop Dance

INTERVENTIONS:
Behavioral: Hip-Hop Dance — I. Week 1 - Session 1
  1. Daily Check-In
  2. Warm-Up: Mobility/Grooves
  3. Lesson: Style - Hip-Hop
  4. Cool-Down: Deep Breathing
  5. Debrief Check-In
  II. Week 2 - Session 2
  1. Daily Check-In
  2. Warm-Up: Mobility/Grooves
  3. Lesson: Style - Locking
  4. Cool-Down: Instructed Yoga
  5. Debrief Check-In
  III. Week 3 - Session 3
  1. Daily Check-In
  2. Warm-Up: Mobility/Grooves
  3. Lesson: Style - Breaking
  4. Cool-Down: Sensory Time
  5. Debrief Check-In
  IV. Week 4 - Session 4
  1. Daily Check-In
  2. Warm-Up: Mobility/Grooves
  3. Lesson: Style - Popping
  4. Cool-Down: Animal Deep Breathing
  5. Debrief Check-In
  V. Week 5 - Session 5
  1. Daily Check-In
  2. Warm-Up: Mobility/Grooves
  3. Lesson: Learn Showcase Routine
  4. Cool-Down: Animal Instructed Yoga
  5. Debrief Check-In
  VI. Week 6 - Session 6
  1. Daily Check-In
  2. Warm-Up: Mobility/Grooves
  3. Lesson: Review Showcase Routine
  4. Cool-Down: Sensory Time
  5. Debrief Check-In
  VII. Week 7 - Dance Showcase

SUMMARY:
This study will explore the effectiveness of dance as an intervention to promote social-emotional health within children with ASD.

DETAILED DESCRIPTION:
The study will look children with ASD's response to a 7-week occupational therapy led dance program in regards to social-emotional health. This will include exploring the effect on change of social-emotional behavior in children with ASD after being exposed to dance intervention through comparing the quantitative measurements of pre- and post-assessment scores of the Developmental Profile 4 (DP-4), analysis of the qualitative measurements of pre- and post-social-emotional behaviors via child report, and analysis of qualitative observations of social-emotional behavior through reviewing video recording of dance classes. Additionally, parents' perspectives will be explored through post-interview questions to share their observations of their child's experience.

ELIGIBILITY:
Inclusion Criteria for Youth Participants

* Elementary school children ages 7-11.
* Parent/caregiver/guardian must provide proof of an Individualized Education Plan (IEP) with a Primary Eligibility of Autism.

  o Parent/caregiver/guardian must provide proof of IEP and eligibility.
* Will speak and understand English.
* Able to physically participate in the dance program without the use of adaptive equipment.
* Answer yes to the following Skillset Checklist (Per parent/caregiver/guardian report):

  * Follow 1- and 2-step instructions.
  * Follow structured activities with supervision (e.g., visual schedule, routine).
  * Previous participation in extracurricular group activities over the last 6 months - 1 year (e.g., structured sports).
  * Minimum 5-minutes of attention to task.

Exclusion Criteria:

* No IEP Primary Eligibility of Autism.
* No children participants younger than 7.
* No children participants older than 11.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2024-05-25 (Actual); Study Completion 2024-05-25 (Actual)

PRIMARY OUTCOMES:
Child Description of Impact on Social-Emotional Health | Change between baseline (time of enrollment) and Week 7
  Subject will be asked to describe emotional state immediately prior to weekly dance intervention and immediately after dance intervention completed. Subject will be asked to verbalize emotional state or choose an icon to represent emotional state. Interviewer will record subject response. Effectiveness will be measured based on verbal or visual responses between 3 options: "Happy", "Sad", or "Okay", where "Happy" is considered effective, "Sad" considered to be ineffective, or if the responses are the same before and after than there is no change. This is a composite measurement over the course of 7 weeks.

SECONDARY OUTCOMES:
Parent Perspective of Impact on Social-Emotional Health | Change between baseline (time of enrollment) and Week 7 (program completion)
  Parent will complete the Developmental Profile 4 (DP-4) assessment pre- and post-program regarding the child's social-emotional behavior. Effectiveness will be measured on responses between "Yes" and "No", where "Yes" is applicable to the parent's child, and "No" is not applicable. This is a composite measurement with 1 domain and 36 sub questions of the assessment before and after the program.
Change in Social-Emotional Behavior | Change between baseline (time of enrollment) and Week 7 (program completion)
  Subjects will be audio/video recorded in each dance class weekly. Researcher will observe and analyze recordings using a developed observation checklist of each subject. Effectiveness will be measured by responses of "Observed" and "Not Observed", where "Observed" is witness in the subject and is effective, and "Not Observed" is not witnessed in the subject and is ineffective.This is a composite measurement over the course of 7 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Loma Linda University Health, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No